CLINICAL TRIAL: NCT06610630
Title: Research on the Application of AI Image Recognition-Based Smartphone Apps in Personalized Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianning Yao (Other)
Responsible Party: Sponsor-Investigator, Jianning Yao, Deputy Chief Physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-KY-1219-001
Record Dates: First submitted 2024-09-21; First posted 2024-09-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Polyps
Keywords: Colonoscopy; bowel preparation; artificial intelligence; smartphone; BBPS score

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted group (Experimental)
  Interventions: Diagnostic Test: Assessment of Bowel Preparation Using AI-Driven Smartphone Applications
- Conventional control group (No Intervention)

INTERVENTIONS:
Diagnostic Test: Assessment of Bowel Preparation Using AI-Driven Smartphone Applications — Assessment of Bowel Preparation Using AI-Driven Smartphone Applications
  Arms: AI-assisted group

SUMMARY:
Colorectal cancer, as one of the most common malignant tumors of the digestive system, has a high incidence and mortality rate worldwide. High-quality colonoscopy is essential for the early detection and prevention of colorectal cancer and is key to improving the survival rates of patients. However, traditional colonoscopy faces numerous challenges in bowel preparation, such as inadequate preparation and a lack of personalized cleansing approaches. Therefore, it is particularly important to develop timely and efficient individualized bowel preparation methods. Artificial intelligence, especially deep learning technologies, has shown great potential in the medical field. This study aims to leverage the advantages of artificial intelligence to optimize the bowel preparation process before colonoscopy, creating a personalized bowel preparation plan that effectively improves the efficacy of colorectal cancer screening and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent painless colonoscopy at the Digestive Endoscopy Center of the First Affiliated Hospital of Zhengzhou University and signed the informed consent for the clinical trial.

Individuals who use smartphones.

Exclusion Criteria:

* Patients with contraindications for colonoscopy. Individuals in whom successful cecal intubation could not be achieved.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | During Colonoscopy
Dosage of Bowel Cleansing Agents | During Bowel Preparation Before Colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No